CLINICAL TRIAL: NCT02758574
Title: Comparison of Standard Catheter Directed Thrombolysis vs. Ultrasound Assisted Thrombolysis for Patients With Acute Submassive Pulmonary Embolism
Brief Title: Standard vs. Ultrasound-assisted Catheter Thrombolysis for Submassive Pulmonary Embolism
Acronym: SUNSET sPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Efthymios Avgerinos, MD, Assistant Professor of Surgery, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO15090058
Record Dates: First submitted 2016-03-22; First posted 2016-05-02 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Embolism
Keywords: acute pulmonary embolism; submassive pulmonary embolism; thrombolysis; catheter directed thrombolysis; ultrasound assisted thrombolysis
MeSH Terms: conditions — Pulmonary Embolism | interventions — carbohydrate-deficient transferrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CDT without ultrasound acceleration (Active Comparator): Standard Catheter-Directed Thrombolysis: Utilization of a standard infusion catheter, placed at the site of pulmonary thrombus. The catheter will be used for the delivery of thrombolytic medications to treat/dissolve pulmonary embolus
  Interventions: Procedure: CDT without ultrasound acceleration
- CDT ultrasound accelerated (Experimental): Ultrasound Accelerated Catheter-Directed Thrombolysis: Utilization of an infusion catheter that incorporates an ultrasound emitting wire both placed at the site of pulmonary thrombus. The catheter will be used for the delivery of thrombolytic medications with the ultrasound emitting wire activated to treat/dissolve pulmonary embolus
  Interventions: Procedure: CDT with ultrasound acceleration

INTERVENTIONS:
Procedure: CDT without ultrasound acceleration — A pulmonary arteriogram will be performed. Upon confirmation of the pulmonary embolus a standard infusion catheter will be placed within the clot. The catheter will be used for infusion of thrombolytics to treat/dissolve the pulmonary embolus.
  Other Names: Standard CDT
  Arms: CDT without ultrasound acceleration
Procedure: CDT with ultrasound acceleration — A pulmonary arteriogram will be performed. Upon confirmation of the pulmonary embolus an infusion catheter that incorporates an ultrasound emitting wire will be placed within the clot. The catheter will be used for infusion of thrombolytics to treat/dissolve the pulmonary embolus. The wire will be connected to an ultrasound generating device.
  Other Names: Ultrasound assisted CDT
  Arms: CDT ultrasound accelerated

SUMMARY:
The study will compare standard catheter directed thrombolysis to ultrasound accelerated thrombolysis for the treatment of acute submassive pulmonary embolism (PE). The study population will include patients eligible for catheter directed thrombolysis (CDT) for submassive PE. Subjects will be randomized to, either, standard catheter-directed thrombolysis or ultrasound-accelerated thrombolysis (USAT).

DETAILED DESCRIPTION:
Acute pulmonary embolism (PE) carries a high morbidity and is the third-leading cause of cardiovascular mortality in the western world. It accounts for 5-10% of in-hospital deaths that for the United States translates to 200,000 deaths per year.1 Recent registries and cohort studies suggest that approximately 10% of all patients with acute PE die during the first 1 to 3 months after diagnosis. Studies that have observed survivors for >3 months have reported an incidence of chronic thromboembolic pulmonary hypertension (CTEPH) 1-5% within 2-3 years after PE.6-10 It is an incapacitating long-term complication of thromboembolic disease with a negative impact on the patient's quality of life and prognosis.

The management acute PE is mainly guided by the acuity and severity of clinical presentation. Initial systemic anticoagulation (AC) is the standard of care and treatment is escalated based on the clinical presentation and patient characteristics that may stratify them at a higher mortality risk. The goals of therapy are to primarily prevent mortality, and secondarily potentially prevent late onset chronic thromboembolic pulmonary hypertension (CTEPH) and improve quality of life.

Massive PE is defined as PE associated with sustained hemodynamic instability, whereas submassive PE (sPE) is defined as PE without hemodynamic instability but with abnormal right ventricular (RV) function and/or evidence of myocardial necrosis. It is notable that there is ongoing interest to accurately risk stratify sPE to identify the patients who are at increased risk of decompensating and/or dying. Clinical scores, imaging tests and biomarkers are under investigation, yet an ideal prognostic tool is still pending. A novel cardiac biomarker, heart-type fatty acid-binding protein (h-FABP), is emerging as a significant predictor of mortality in patients with submassive PE.

Systemic intravenous thrombolysis is universally recommended by all guideline bodies for massive pulmonary embolism, but remains controversial for submassive PE. In the most recent metaanalysis, the subgroup analysis of 8 submassive PE trials (1993-2014, n=1775) showed that thrombolytic therapy was associated with a mortality reduction (1.39% vs 2.92%) but with an increase in major bleeding (7.74% vs 2.25%). These results were mainly driven by the largest randomized trial (PEITHO, 1006 patients) which compared a single, weight-adapted i.v. bolus of tenecteplase with standard anticoagulation.

The recent development of catheter-directed therapies such as catheter-directed thrombolysis (CDT), ultrasound-accelerated thrombolysis (USAT), and pharmacomechanical or aspiration thrombectomy has introduced more tools for the treatment of acute PE. Proponents of these techniques suggest that they may provide a similar therapeutic benefit as systemic thrombolysis, while decreasing the dose of thrombolytic required and potentially decreasing the risk of adverse bleeding events. Both the American Heart Association and more recently European Society of Cardiology have acknowledged CDT as a viable treatment alternative for high risk acute sPE (echocardiographic RV dysfunction and elevated cardiac biomarkers), if appropriate expertise is available and particularly when the bleeding risk is high.

Catheter-directed thrombolysis requires placement of a multi-sidehole infusion catheter within the pulmonary arterial thrombus burden under angiographic guidance. Thrombolytic medications are slowly infused through the catheter, which is left in place for the duration of the treatment. USAT is a modification of this therapy utilizing a proprietary system of local high frequency, low-power ultrasound to dissociate the fibrin matrix of the thrombus, allowing deeper penetration of lytic medication.

Several observational non-controlled series have demonstrated the efficacy of catheter-directed techniques in improving clinical and hemodynamic parameters and reducing clot burden while demonstrating a favorable safety profile. The ULTIMA trial was the first randomized controlled trial to include CDIs for sPE comparing standardized fixed-dose of USAT (10mg rtPA per lung over 15 hours) and AC to AC alone. In the USAT group, but not in the heparin group, the mean RV/LV ratio was significantly reduced at 24 hours, but became comparable between the two groups at 90 days. The RV systolic function was significantly improved in the USAT group vs. the heparin group at both 24 hours and 90 days. In both study groups minor bleeding complications were rare and there were no major bleeding complications. The SEATTLE II trial, a single-arm study evaluating the effectiveness of USAT, showed also an RV/LV ratio improvement at 48 hours.

Limited data exists for comparing different catheter-directed therapies for acute PE. The majority of recent series for catheter-directed interventions utilize USAT exclusively; however there is limited comparative effectiveness data comparing this modality to standard multi-sidehole catheter infusion. Preliminary, non-controlled data are conflicting. One series by Lin and colleagues of 33 high-risk PE patients suggested benefit for USAT for angiographic clearance of thrombus burden with more bleeding events in the CDT group.31 Kuo and colleagues noted no difference in outcomes and treatment specifics between USAT and CDT in the recently published early results of a multicenter prospective registry. Our retrospective analysis of 63 patients suggests that there may be no difference between the two treatment modalities, demonstrating similar rates of outcomes such as survival, hemodynamic stabilization, and echocardiographic parameters in both groups with similar procedure length and lytic dose in the time-adjusted cohorts. Selection bias cannot be underestimated in all these studies.

The expected benefit of USAT has been dependent on the device's ability to increase penetration of lytic into thrombus using high frequency, low power ultrasound, due to its reversible effects on fibrin dissociation. This benefit has been shown to result in faster thrombus clearance in selected vascular beds in some studies, such as the recently published DUET study comparing USAT and CDT in arterial occlusions. More rapid clearance of pulmonary thrombus by USAT compared to standard CDT may prove to be clinically and cost effective (e.g. via reduced length of ICU and hospital stay). Alternatively, if thrombus clearance is similar, the cost of USAT may exceed the cost of CDT (proprietary equipment and disposables), without offering any potential advantage. Evidence from the venous circulation, coming from the recent BERNUTIFUL trial demonstrated no difference in time to thrombus clearance in lower extremity deep venous thrombosis.

ELIGIBILITY:
Criteria: Inclusion Criteria:

* Subject is eligible for catheter directed thrombolysis per the study protocol for submassive PE (CT or echocardiographic RV strain (defined as RV/LV ratio >1) without persisting hypotension <90mmHg or drop of systolic blood pressure by at least 40mm Hg for at least 15 minutes with signs of end-organ hypoperfusion (cold extremities or low urinary output <30 mL/h or mental confusion) and without the need of catecholamine support or cardiopulmonary resuscitation).

Exclusion Criteria:

* pregnancy;
* index PE symptom duration >14 days;
* high bleeding rsk (any prior intracranial hemorrhage,
* known structural intracranial cerebrovascular disease or neoplasm,
* ischemic stroke within 3 months,
* suspected aortic dissection, active bleeding or bleeding diathesis,
* recent spinal or cranial/brain surgery,
* recent closed-head or facial trauma with bony fracture or brain injury);
* participation in any other investigational drug or device study;
* life expectancy <90 days;
* inability to comply with study assessments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-05; Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
PE thrombus load reduction (CT obstruction index) from baseline to the termination of lysis | 48 hours

SECONDARY OUTCOMES:
Mortality | 90 days
Stroke | 30 days
  Any ischemic or hemorrhagic stroke
Major Bleeding | 30 days
  Any major bleeding event defined as hemorrhagic stroke, need to transfuse or need to intervene
Echocardiographic Right Ventricular/Left Ventricular Diameter (ratio) | 12 months
Functional status (6 min walk test) | 12 months
  6 min walk test (meters)
Cost effectiveness analysis | 12 months
  Quality Adjusted Life Years - Costs based on in-hospital resource utilization and out-of hospital care and follow-up.
Echocardiographic Tricuspid Annular Plane Systolic Excursion (cm) | 12 months
Quality of life Questionnaire SF36 (score) | 12 months
Quality of life Questionnaire PE QOL (score) | 12 months
Quality of life Questionnaire San Diego Shortness of Breath (score) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Efthymios Avgerinos, M.D., Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC Mercy, Pittsburgh, Pennsylvania
  - UPMC Shadyside, Pittsburgh, Pennsylvania
  - UPMC Passavant, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kahn SR, Houweling AH, Granton J, Rudski L, Dennie C, Hirsch A. Long-term outcomes after pulmonary embolism: current knowledge and future research. Blood Coagul Fibrinolysis. 2014 Jul;25(5):407-15. doi: 10.1097/MBC.0000000000000070. PMID 24469387
- [Background] Avgerinos ED, Chaer RA. Catheter-directed interventions for acute pulmonary embolism. J Vasc Surg. 2015 Feb;61(2):559-65. doi: 10.1016/j.jvs.2014.10.036. Epub 2014 Dec 16. PMID 25524824
- [Background] Jaff MR, McMurtry MS, Archer SL, Cushman M, Goldenberg N, Goldhaber SZ, Jenkins JS, Kline JA, Michaels AD, Thistlethwaite P, Vedantham S, White RJ, Zierler BK; American Heart Association Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation; American Heart Association Council on Peripheral Vascular Disease; American Heart Association Council on Arteriosclerosis, Thrombosis and Vascular Biology. Management of massive and submassive pulmonary embolism, iliofemoral deep vein thrombosis, and chronic thromboembolic pulmonary hypertension: a scientific statement from the American Heart Association. Circulation. 2011 Apr 26;123(16):1788-830. doi: 10.1161/CIR.0b013e318214914f. Epub 2011 Mar 21. PMID 21422387
- [Background] Kearon C, Akl EA, Comerota AJ, Prandoni P, Bounameaux H, Goldhaber SZ, Nelson ME, Wells PS, Gould MK, Dentali F, Crowther M, Kahn SR. Antithrombotic therapy for VTE disease: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e419S-e496S. doi: 10.1378/chest.11-2301. PMID 22315268
- [Background] Konstantinides SV, Torbicki A, Agnelli G, Danchin N, Fitzmaurice D, Galie N, Gibbs JS, Huisman MV, Humbert M, Kucher N, Lang I, Lankeit M, Lekakis J, Maack C, Mayer E, Meneveau N, Perrier A, Pruszczyk P, Rasmussen LH, Schindler TH, Svitil P, Vonk Noordegraaf A, Zamorano JL, Zompatori M; Task Force for the Diagnosis and Management of Acute Pulmonary Embolism of the European Society of Cardiology (ESC). 2014 ESC guidelines on the diagnosis and management of acute pulmonary embolism. Eur Heart J. 2014 Nov 14;35(43):3033-69, 3069a-3069k. doi: 10.1093/eurheartj/ehu283. Epub 2014 Aug 29. No abstract available. PMID 25173341
- [Background] Becattini C, Agnelli G, Pesavento R, Silingardi M, Poggio R, Taliani MR, Ageno W. Incidence of chronic thromboembolic pulmonary hypertension after a first episode of pulmonary embolism. Chest. 2006 Jul;130(1):172-5. doi: 10.1378/chest.130.1.172. PMID 16840398
- [Background] Meyer G, Planquette B, Sanchez O. Long-term outcome of pulmonary embolism. Curr Opin Hematol. 2008 Sep;15(5):499-503. doi: 10.1097/MOH.0b013e3283063a51. PMID 18695374
- [Background] Pengo V, Lensing AW, Prins MH, Marchiori A, Davidson BL, Tiozzo F, Albanese P, Biasiolo A, Pegoraro C, Iliceto S, Prandoni P; Thromboembolic Pulmonary Hypertension Study Group. Incidence of chronic thromboembolic pulmonary hypertension after pulmonary embolism. N Engl J Med. 2004 May 27;350(22):2257-64. doi: 10.1056/NEJMoa032274. PMID 15163775
- [Background] Sanchez O, Trinquart L, Colombet I, Durieux P, Huisman MV, Chatellier G, Meyer G. Prognostic value of right ventricular dysfunction in patients with haemodynamically stable pulmonary embolism: a systematic review. Eur Heart J. 2008 Jun;29(12):1569-77. doi: 10.1093/eurheartj/ehn208. Epub 2008 May 21. PMID 18495689
- [Background] Guerin L, Couturaud F, Parent F, Revel MP, Gillaizeau F, Planquette B, Pontal D, Guegan M, Simonneau G, Meyer G, Sanchez O. Prevalence of chronic thromboembolic pulmonary hypertension after acute pulmonary embolism. Prevalence of CTEPH after pulmonary embolism. Thromb Haemost. 2014 Sep 2;112(3):598-605. doi: 10.1160/TH13-07-0538. Epub 2014 Jun 5. PMID 24898545
- [Background] Chatterjee S, Chakraborty A, Weinberg I, Kadakia M, Wilensky RL, Sardar P, Kumbhani DJ, Mukherjee D, Jaff MR, Giri J. Thrombolysis for pulmonary embolism and risk of all-cause mortality, major bleeding, and intracranial hemorrhage: a meta-analysis. JAMA. 2014 Jun 18;311(23):2414-21. doi: 10.1001/jama.2014.5990. PMID 24938564
- [Background] Fasullo S, Scalzo S, Maringhini G, Ganci F, Cannizzaro S, Basile I, Cangemi D, Terrazzino G, Parrinello G, Sarullo FM, Baglini R, Paterna S, Di Pasquale P. Six-month echocardiographic study in patients with submassive pulmonary embolism and right ventricle dysfunction: comparison of thrombolysis with heparin. Am J Med Sci. 2011 Jan;341(1):33-9. doi: 10.1097/MAJ.0b013e3181f1fc3e. PMID 20890176
- [Background] Kline JA, Steuerwald MT, Marchick MR, Hernandez-Nino J, Rose GA. Prospective evaluation of right ventricular function and functional status 6 months after acute submassive pulmonary embolism: frequency of persistent or subsequent elevation in estimated pulmonary artery pressure. Chest. 2009 Nov;136(5):1202-1210. doi: 10.1378/chest.08-2988. Epub 2009 Jun 19. PMID 19542256
- [Background] Sharifi M, Bay C, Skrocki L, Rahimi F, Mehdipour M; "MOPETT" Investigators. Moderate pulmonary embolism treated with thrombolysis (from the "MOPETT" Trial). Am J Cardiol. 2013 Jan 15;111(2):273-7. doi: 10.1016/j.amjcard.2012.09.027. Epub 2012 Oct 24. PMID 23102885
- [Background] Ain DL, Jaff MR. Treatment of Submassive Pulmonary Embolism: Knowing When to be Aggressive and When to be Conservative. Curr Treat Options Cardiovasc Med. 2015 Jun;17(6):385. doi: 10.1007/s11936-015-0385-y. PMID 25895738
- [Background] Klok FA, Meyer G, Konstantinides S. Management of intermediate-risk pulmonary embolism: uncertainties and challenges. Eur J Haematol. 2015 Dec;95(6):489-97. doi: 10.1111/ejh.12612. Epub 2015 Jul 15. PMID 26109174
- [Background] Weinberg I, Jaff MR. Treating large pulmonary emboli: do the guidelines guide us? Curr Opin Pulm Med. 2013 Sep;19(5):413-21. doi: 10.1097/MCP.0b013e3283642a63. PMID 23884294
- [Background] Meyer G, Vicaut E, Danays T, Agnelli G, Becattini C, Beyer-Westendorf J, Bluhmki E, Bouvaist H, Brenner B, Couturaud F, Dellas C, Empen K, Franca A, Galie N, Geibel A, Goldhaber SZ, Jimenez D, Kozak M, Kupatt C, Kucher N, Lang IM, Lankeit M, Meneveau N, Pacouret G, Palazzini M, Petris A, Pruszczyk P, Rugolotto M, Salvi A, Schellong S, Sebbane M, Sobkowicz B, Stefanovic BS, Thiele H, Torbicki A, Verschuren F, Konstantinides SV; PEITHO Investigators. Fibrinolysis for patients with intermediate-risk pulmonary embolism. N Engl J Med. 2014 Apr 10;370(15):1402-11. doi: 10.1056/NEJMoa1302097. PMID 24716681
- [Background] Engelberger RP, Kucher N. Ultrasound-assisted thrombolysis for acute pulmonary embolism: a systematic review. Eur Heart J. 2014 Mar;35(12):758-64. doi: 10.1093/eurheartj/ehu029. Epub 2014 Feb 3. PMID 24497337
- [Background] Engelhardt TC, Taylor AJ, Simprini LA, Kucher N. Catheter-directed ultrasound-accelerated thrombolysis for the treatment of acute pulmonary embolism. Thromb Res. 2011 Aug;128(2):149-54. doi: 10.1016/j.thromres.2011.05.014. Epub 2011 Jun 8. PMID 21641020
- [Background] Kucher N, Boekstegers P, Muller OJ, Kupatt C, Beyer-Westendorf J, Heitzer T, Tebbe U, Horstkotte J, Muller R, Blessing E, Greif M, Lange P, Hoffmann RT, Werth S, Barmeyer A, Hartel D, Grunwald H, Empen K, Baumgartner I. Randomized, controlled trial of ultrasound-assisted catheter-directed thrombolysis for acute intermediate-risk pulmonary embolism. Circulation. 2014 Jan 28;129(4):479-86. doi: 10.1161/CIRCULATIONAHA.113.005544. Epub 2013 Nov 13. PMID 24226805
- [Background] Kuo WT. Endovascular therapy for acute pulmonary embolism. J Vasc Interv Radiol. 2012 Feb;23(2):167-79.e4; quiz 179. doi: 10.1016/j.jvir.2011.10.012. Epub 2011 Dec 20. PMID 22192633
- [Background] Kuo WT, Gould MK, Louie JD, Rosenberg JK, Sze DY, Hofmann LV. Catheter-directed therapy for the treatment of massive pulmonary embolism: systematic review and meta-analysis of modern techniques. J Vasc Interv Radiol. 2009 Nov;20(11):1431-40. doi: 10.1016/j.jvir.2009.08.002. PMID 19875060
- [Background] Weinberg I, Jaff MR. Accelerated thrombolysis for pulmonary embolism: will clinical benefit be ULTIMAtely realized? Circulation. 2014 Jan 28;129(4):420-1. doi: 10.1161/CIRCULATIONAHA.113.007132. Epub 2013 Nov 13. No abstract available. PMID 24226804
- [Background] Bagla S, Smirniotopoulos JB, van Breda A, Sheridan MJ, Sterling KM. Ultrasound-accelerated catheter-directed thrombolysis for acute submassive pulmonary embolism. J Vasc Interv Radiol. 2015 Jul;26(7):1001-6. doi: 10.1016/j.jvir.2014.12.017. Epub 2015 Feb 18. PMID 25704224
- [Background] George B, Wallace EL, Charnigo R, Wingerter KE, Kapadia P, Gurley JC, Smyth SS. A retrospective analysis of catheter-based thrombolytic therapy for acute submassive and massive pulmonary embolism. Vasc Med. 2015 Apr;20(2):122-30. doi: 10.1177/1358863X14568135. PMID 25832600
- [Background] McCabe JM, Huang PH, Riedl L, Eisenhauer AC, Sobieszczyk P. Usefulness and safety of ultrasound-assisted catheter-directed thrombolysis for submassive pulmonary emboli. Am J Cardiol. 2015 Mar 15;115(6):821-4. doi: 10.1016/j.amjcard.2014.12.050. Epub 2015 Jan 7. PMID 25633189
- [Background] Kuo WT, Banerjee A, Kim PS, DeMarco FJ Jr, Levy JR, Facchini FR, Unver K, Bertini MJ, Sista AK, Hall MJ, Rosenberg JK, De Gregorio MA. Pulmonary Embolism Response to Fragmentation, Embolectomy, and Catheter Thrombolysis (PERFECT): Initial Results From a Prospective Multicenter Registry. Chest. 2015 Sep;148(3):667-673. doi: 10.1378/chest.15-0119. PMID 25856269
- [Background] Piazza G ET, Sterling KM, et al. A prospective, single-arm, multicenter trial of the ekosonic endovascular system with activase for acute pulmonary embolism (seattle II). American College of Cardiology 63rd Annual Scientific Meeting. 2014
- [Background] Warntges S, Konstantinides SV. Progress in the management of acute pulmonary embolism. Curr Opin Pulm Med. 2015 Sep;21(5):417-24. doi: 10.1097/MCP.0000000000000196. PMID 26186247
- [Background] Lin PH, Annambhotla S, Bechara CF, Athamneh H, Weakley SM, Kobayashi K, Kougias P. Comparison of percutaneous ultrasound-accelerated thrombolysis versus catheter-directed thrombolysis in patients with acute massive pulmonary embolism. Vascular. 2009 Nov-Dec;17 Suppl 3:S137-47. doi: 10.2310/6670.2009.00063. PMID 19919804
- [Background] Liang NL, Avgerinos ED, Marone LK, Singh MJ, Makaroun MS, Chaer RA. Equivalent Outcomes Between Ultrasound-Assisted Thrombolysis and Standard Catheter-Directed Thrombolysis for the Treatment of Acute Pulmonary Embolism. J Vasc Surg Venous Lymphat Disord. 2015 Jan;3(1):120-1. doi: 10.1016/j.jvsv.2014.10.015. Epub 2014 Dec 15. No abstract available. PMID 26993702
- [Background] Schrijver AM, van Leersum M, Fioole B, Reijnen MM, Hoksbergen AW, Vahl AC, de Vries JP. Dutch randomized trial comparing standard catheter-directed thrombolysis and ultrasound-accelerated thrombolysis for arterial thromboembolic infrainguinal disease (DUET). J Endovasc Ther. 2015 Feb;22(1):87-95. doi: 10.1177/1526602814566578. PMID 25775686
- [Background] Engelberger RP, Spirk D, Willenberg T, Alatri A, Do DD, Baumgartner I, Kucher N. Ultrasound-assisted versus conventional catheter-directed thrombolysis for acute iliofemoral deep vein thrombosis. Circ Cardiovasc Interv. 2015 Jan;8(1):e002027. doi: 10.1161/CIRCINTERVENTIONS.114.002027. PMID 25593121
- [Background] Qanadli SD, El Hajjam M, Vieillard-Baron A, Joseph T, Mesurolle B, Oliva VL, Barre O, Bruckert F, Dubourg O, Lacombe P. New CT index to quantify arterial obstruction in pulmonary embolism: comparison with angiographic index and echocardiography. AJR Am J Roentgenol. 2001 Jun;176(6):1415-20. doi: 10.2214/ajr.176.6.1761415. PMID 11373204
- [Background] Mastora I, Remy-Jardin M, Masson P, Galland E, Delannoy V, Bauchart JJ, Remy J. Severity of acute pulmonary embolism: evaluation of a new spiral CT angiographic score in correlation with echocardiographic data. Eur Radiol. 2003 Jan;13(1):29-35. doi: 10.1007/s00330-002-1515-y. Epub 2002 Jun 19. PMID 12541107
- [Background] Gorkin L, Norvell NK, Rosen RC, Charles E, Shumaker SA, McIntyre KM, Capone RJ, Kostis J, Niaura R, Woods P, et al. Assessment of quality of life as observed from the baseline data of the Studies of Left Ventricular Dysfunction (SOLVD) trial quality-of-life substudy. Am J Cardiol. 1993 May 1;71(12):1069-73. doi: 10.1016/0002-9149(93)90575-w. PMID 8475871
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Kennedy RJ, Kenney HH, Dunfee BL. Thrombus resolution and hemodynamic recovery using ultrasound-accelerated thrombolysis in acute pulmonary embolism. J Vasc Interv Radiol. 2013 Jun;24(6):841-8. doi: 10.1016/j.jvir.2013.02.023. Epub 2013 Apr 16. PMID 23601295
- [Background] Blinc A, Francis CW, Trudnowski JL, Carstensen EL. Characterization of ultrasound-potentiated fibrinolysis in vitro. Blood. 1993 May 15;81(10):2636-43. PMID 8490172
- [Background] Francis CW, Blinc A, Lee S, Cox C. Ultrasound accelerates transport of recombinant tissue plasminogen activator into clots. Ultrasound Med Biol. 1995;21(3):419-24. doi: 10.1016/0301-5629(94)00119-x. PMID 7645133
- [Derived] Andraska EA, Bonaroti J, Zhang Y, Rivera-Lebron B, Chaer RA, Avgerinos ED. Predictors of chronic thromboembolic pulmonary hypertension in patients with submassive pulmonary embolism treated with catheter-directed thrombolysis versus anticoagulation alone: A secondary analysis of the SUNSET sPE trial. J Vasc Surg Venous Lymphat Disord. 2023 Nov;11(6):1157-1164. doi: 10.1016/j.jvsv.2023.06.003. Epub 2023 Jun 22. PMID 37353154
- [Derived] Avgerinos ED, Mohapatra A, Rivera-Lebron B, Toma C, Kabrhel C, Fish L, Lacomis J, Ocak I, Chaer RA; PERT Consortium. Design and rationale of a randomized trial comparing standard versus ultrasound-assisted thrombolysis for submassive pulmonary embolism. J Vasc Surg Venous Lymphat Disord. 2018 Jan;6(1):126-132. doi: 10.1016/j.jvsv.2017.09.004. PMID 29248101